CLINICAL TRIAL: NCT03626883
Title: Single Versus Double Hamstring Harvest for Anterior Cruciate Ligament Reconstruction. Clinical, Laboratory, Radiographic and Patient-reported Outcomes
Brief Title: Single Versus Double Hamstring Harvest for Anterior Cruciate Ligament Reconstruction
Acronym: 1vs2ham
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rafał Kamiński (Other)
Responsible Party: Sponsor-Investigator, Rafał Kamiński, MD, PhD, Centre of Postgraduate Medical Education
Organization: Centre of Postgraduate Medical Education (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1vs2 ham
Record Dates: First submitted 2018-02-13; First posted 2018-08-13 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: arthroscopy
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 hamstring (Experimental): Patients will receive the intervention of 'single-bundle, single-hamstring ACL reconstruction'.
  Interventions: Procedure: single-bundle, single-hamstring ACL reconstruction
- 2 hamstrings (Active Comparator): Patients will receive the intervention of 'single-bundle, double-hamstring ACL reconstruction'.
  Interventions: Procedure: single-bundle, double-hamstring ACL reconstruction

INTERVENTIONS:
Procedure: single-bundle, single-hamstring ACL reconstruction — anterior cruciate ligament reconstruction with single hamstring tendon
  Arms: 1 hamstring
Procedure: single-bundle, double-hamstring ACL reconstruction — anterior cruciate ligament reconstruction with 2 hamstring tendons
  Arms: 2 hamstrings

SUMMARY:
The aim of the study is to examine the influence of number of the harvested hamstring tendons on subjective and objective outcomes of primary anterior cruciate ligament reconstruction.

DETAILED DESCRIPTION:
The aim of the study is to examine the influence of number of the harvested hamstring tendons on subjective (patient-reported outcome measures) and objective (instrument-tested and imaging studies) outcomes of primary anterior cruciate ligament reconstruction.

The study will recruit 60 patients per each of two arms.

ELIGIBILITY:
Inclusion Criteria:

* chronic anterior knee instability with MRI-confirmed anterior cruciate ligament tear

Exclusion Criteria:

* revision anterior cruciate ligament surgery
* other lower limb injuries

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Knee stability (KT1000 assessment), pivot shift at 2,4 and 5yrs time-points | up to 5yrs

SECONDARY OUTCOMES:
Change from baseline International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Form at 104 weeks | up to 5yrs
  Anderson, AF. Rating scales. In: Fu, FH.; Harner, CD.; Vince, KL., editors. Knee surgery.
  Baltimore: Williams & Wilkins; 1994. p. 275-96.
Change from baseline Knee injury and Osteoarthritis Outcome Score at up to 5yrs | up to 5yrs
  Knee injury and Osteoarthritis Outcome Score minimum score:0, maximum score:100 Baltimore: Williams & Wilkins; 1994. p. 275-96.
Change from baseline Lysholm Knee Questionnaire at 104 weeks | up to 5yrs
  Knee function questionnaire (patient-administered), minimum score: 0, maximum score: 100. Full description in: Lysholm J, Gillquist J. Evaluation of knee ligament surgery results with special emphasis on use of a scoring scale. Am J Sports Med. 1982; 10:150-4. [PubMed: 6896798]
Change from baseline Visual Analog Scale for Pain at 104 weeks | up to 5yrs
  Separate Outcome Measure, with minimum 0 and maximum of 10. Full description in: Hawker GA, Mian S, Kendzerska T, French M. Measures of adult pain: Visual Analog Scale for Pain (VAS Pain), Numeric Rating Scale for Pain (NRS Pain), McGill Pain Questionnaire (MPQ), Short-Form McGill Pain Questionnaire (SF-MPQ), Chronic Pain Grade Scale (CPGS), Short Form-36 Bodily Pain Scale (SF-36 BPS), and Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP).
  Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S240-52. doi:10.1002/acr.20543.
Change from baseline tunnel volume at 104 weeks | 104-weeks postop
  Change from baseline tunnel volume will be calculated on magnetic resonance imaging images at 104 weeks postoperatively
Change from baseline tunnel diameter at 104 weeks | 104-weeks postop
  Change from baseline tunnel diameter will be calculated on standing knee x-rays at 104 weeks postoperatively
Need for arthrocentesis, revision surgery, additional procedures up to 104 weeks | up to 5yrs
  The medical records will be prospectively abstracted and analyzed for any arthrocentesis, revision surgery or additional procedures performed in the study group up top 104 weeks after index surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin K Wasko, M.D., Ph.D., Principal Investigator — Centre for Postgraduate Medical Education in Warsaw
Locations (1):
- Prof. A. Gruca Teaching Hospital, Centre for Postgraduate Medical Education, Otwock, Woj. Mazowieckie, Poland

REFERENCES:
- [Derived] Kulinski K, Wasko MK, Trams E, Malesa K, Pomianowski S, Kaminski R. Anterior Cruciate Ligament Reconstruction Using a 4-Strand Semitendinosus Tendon Graft or a Doubled Semitendinosus and Gracilis Tendon Graft: A 4.5-Year Prospective, Randomized, Double-Blind, Parallel-Group Study. Am J Sports Med. 2023 Mar;51(3):615-626. doi: 10.1177/03635465221149738. PMID 36856280